CLINICAL TRIAL: NCT03489187
Title: Visualase Visualization Database (VIVID-1)
Acronym: VIVID-1
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17033NS
Record Dates: First submitted 2018-01-18; First posted 2018-04-05 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy; Tumor; Other
MeSH Terms: conditions — Epilepsy; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- VTTS as standard of care: VTTS as standard of care.
  Interventions: Device: Visualase Thermal Therapy System

INTERVENTIONS:
Device: Visualase Thermal Therapy System — Patients who have previously received treatment with VTTS when used as intended.
  Other Names: VTTS

SUMMARY:
The purpose of the VIVID-1 data collection study is to establish a database of clinical images and associated technical files from commercial cases using the Visualase Thermal Therapy System (VTTS). All data collected will be de-identified. No safety or effectiveness assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient correlating with the de-identified data set to be collected received standard of care treatment using the Visualase System prior to the date of site activation.

Exclusion Criteria:

1. Patient correlating with the de-identified data set to be collected is a minor (less than 18 years old, or as defined by local policy) that is not allowed to participate in this type of research project (eg, IRB approval with waiver of consent) per IRB policy
2. Patient correlating with the de-identified data set to be collected is enrolled in the Medtronic SLATE trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have previously received treatment with VTTS when used as intended.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Image assessment | During the Procedure
  Identify pathologies and tissue types prescribed Visualse Thermal Therapy

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Rutgers, New Brunswick, New Jersey
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - University of Washington Harborview, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No